CLINICAL TRIAL: NCT02682706
Title: Magnetic Resonance Imaging of Human Supraclavicular Brown Adipose Tissue - MIBAT Study
Acronym: MIBAT
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EKNZ BASEC 2015-00199
Record Dates: First submitted 2016-02-10; First posted 2016-02-15 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Healthy
Keywords: brown adipose tissue; magnetic resonance imaging; energy expenditure; non-shivering thermogenesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Brown adipose tissue (BAT) is unique in its capability to convert chemical energy directly into heat. Active BAT increases energy expenditure and can thereby counteract obesity and insulin resistance. Currently, the imaging method of choice to assess BAT morphology and function is 18F-FDG-PET/CT which is expensive and exposes patients or healthy volunteers to ionizing radiation, thus impeding larger prospective studies.

Magnetic resonance imaging (MRI) could constitute a suitable alternative and preliminary small-scale studies are promising.

The overall aim of this research proposal is to develop reliable magnetic resonance imaging techniques to facilitate the study of brown adipose tissue in human adults, specifically in the context of endocrine disease.

Specifically, investigators want to

1. Develop a reliable MR imaging protocol for human BAT and compare BAT volume to cold induced nonshivering thermogenesis as a measure of BAT activity.
2. Assess the intra-individual variance of BAT volume measured by MRI.
3. Evaluate direct measurement of BAT temperature by functional MRI.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age 18-40 years
* Body mass index (BMI): 17.5-27 kg/m²

Exclusion Criteria:

* known concomitant disease influencing thyroid hormone metabolism
* severe diseases: chronic heart failure, liver cirrhosis, kidney failure, active cancer
* known hypersensitivity to cold, e.g. primary or secondary Raynaud's syndrome
* abuse of alcohol or illicit drugs
* Women who are pregnant or breast feeding
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Previous enrolment into the current study
* implanted device not compatible with MRI, e.g. pace maker

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Correlation of scBAT volume and cold induced thermogenesis as determined by indirect calorimetry | both measurements within 2 weeks
  measurement of scBAT volume and measurement of cold induced thermogenesis as determined by indirect calorimetry, both values measured in a timeframe of two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthias J Betz, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Department of Endocrinology, Basel, Canton of Basel-City
  - University Hospital of Basel, Department of Radiology, Basel, Canton of Basel-City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Senn JR, Maushart CI, Gashi G, Michel R, Lalive d'Epinay M, Vogt R, Becker AS, Muller J, Balaz M, Wolfrum C, Burger IA, Betz MJ. Outdoor Temperature Influences Cold Induced Thermogenesis in Humans. Front Physiol. 2018 Aug 23;9:1184. doi: 10.3389/fphys.2018.01184. eCollection 2018. PMID 30190681